CLINICAL TRIAL: NCT05465499
Title: Preliminary Survey in Preparation for the Implementation of ERAS at Dr Soetomo Hospital
Status: Completed | Type: Observational
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Anna Surgean Veterini, dr., SpAn., KIC, Head of Anesthesiology and Reanimation Installation ; Principal Investigator, Dr. Soetomo General Hospital
Other Study IDs: 0815/LOE/301.4.2/III/2022
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: ERAS
Keywords: ERAS; Intraoperative care; Perioperative care; Preoperative care; Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient: Patient baseline data were taken from the examination at the anesthesiology outpatient clinic. (N=41)
  Interventions: Procedure: ERAS
- Doctor: Consists of specialist and resident anesthesiology, orthopaedic surgery and traumatology, obstetrics and gynaecology, urology. (N=110)
- Healthcare worker: Consists of nutritionists, pharmacists, surgical nurses, anesthesiologists, and recovery room nurses.(N=56)

INTERVENTIONS:
Procedure: ERAS — This study is a cross-sectional observational study by distributing questionnaires regarding the readiness to implement ERAS at Dr Soetomo General Hospital to the subjects, so there is no treatment whatsoever on the subjects.
  Groups: Patient

SUMMARY:
This study aims to analyze the readiness of the team that will support the ERAS application at Regional General Academic Hospital Dr Soetomo.

DETAILED DESCRIPTION:
This is an observational analytic study with a cross-sectional design using a questionnaire. Patient baseline data were taken from the examination at the anesthesiology outpatient clinic. The patient's level of understanding was assessed by two investigators and rated on a scale of 1 to 5. Primary data and assessment of understanding of doctors and medical personnel were filled in independently by research subjects on online forms and rated on a scale of 1 to 5.

ELIGIBILITY:
Inclusion Criteria:

* Patients with elective cesarean, urology, and simple orthopaedic surgery plans
* Patient with PS ASA 1-2

Exclusion Criteria:

* Patients with communication disorders / mental disorders
* Patients with outpatient surgery plans

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who come to the anesthesiology polyclinic to prepare for SC surgery, simple urology, and simple orthopaedics.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Level of understanding (using questionnaire) | 1 month
  This outcome is reported by a score on a scale. The minimum value is one, and the maximum value is five. Higher scores mean better outcomes.
  Scale title:
  1. Strongly don't understand
  2. Don't understand
  3. Neutral
  4. Understand
  5. Strongly understand

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD able to be shared with other researchers with permission

REFERENCES:
- [Background] Pache B, Hübner M, Martin D, Addor V, Ljungqvist O, Demartines N, et al. Requirements for a successful Enhanced Recovery After Surgery (ERAS) program: a multicenter international survey among ERAS nurses. Eur Surg - Acta Chir Austriaca 2021;53:246-50. https://doi.org/10.1007/s10353-021-00698-9.
- [Background] Pedziwiatr M, Kisialeuski M, Wierdak M, Stanek M, Natkaniec M, Matlok M, Major P, Malczak P, Budzynski A. Early implementation of Enhanced Recovery After Surgery (ERAS(R)) protocol - Compliance improves outcomes: A prospective cohort study. Int J Surg. 2015 Sep;21:75-81. doi: 10.1016/j.ijsu.2015.06.087. Epub 2015 Jul 29. PMID 26231994
- [Background] Feldheiser A, Aziz O, Baldini G, Cox BP, Fearon KC, Feldman LS, Gan TJ, Kennedy RH, Ljungqvist O, Lobo DN, Miller T, Radtke FF, Ruiz Garces T, Schricker T, Scott MJ, Thacker JK, Ytrebo LM, Carli F. Enhanced Recovery After Surgery (ERAS) for gastrointestinal surgery, part 2: consensus statement for anaesthesia practice. Acta Anaesthesiol Scand. 2016 Mar;60(3):289-334. doi: 10.1111/aas.12651. Epub 2015 Oct 30. PMID 26514824
- [Background] Geltzeiler CB, Rotramel A, Wilson C, Deng L, Whiteford MH, Frankhouse J. Prospective study of colorectal enhanced recovery after surgery in a community hospital. JAMA Surg. 2014 Sep;149(9):955-61. doi: 10.1001/jamasurg.2014.675. PMID 25054315
- [Background] Melnyk M, Casey RG, Black P, Koupparis AJ. Enhanced recovery after surgery (ERAS) protocols: Time to change practice? Can Urol Assoc J. 2011 Oct;5(5):342-8. doi: 10.5489/cuaj.11002. PMID 22031616
- [Background] Abeles A, Kwasnicki RM, Darzi A. Enhanced recovery after surgery: Current research insights and future direction. World J Gastrointest Surg. 2017 Feb 27;9(2):37-45. doi: 10.4240/wjgs.v9.i2.37. PMID 28289508
- [Background] Springer JE, Doumouras AG, Lethbridge S, Forbes S, Eskicioglu C. A Provincial Assessment of the Barriers and Utilization of Enhanced Recovery After Colorectal Surgery. J Surg Res. 2019 Mar;235:521-528. doi: 10.1016/j.jss.2018.10.047. Epub 2018 Nov 26. PMID 30691838
- [Background] Wang D, Liu Z, Zhou J, Yang J, Chen X, Chang C, Liu C, Li K, Hu J. Barriers to implementation of enhanced recovery after surgery (ERAS) by a multidisciplinary team in China: a multicentre qualitative study. BMJ Open. 2022 Mar 14;12(3):e053687. doi: 10.1136/bmjopen-2021-053687. PMID 35288383
- [Background] Polle SW, Wind J, Fuhring JW, Hofland J, Gouma DJ, Bemelman WA. Implementation of a fast-track perioperative care program: what are the difficulties? Dig Surg. 2007;24(6):441-9. doi: 10.1159/000108327. Epub 2007 Sep 13. PMID 17851238
- [Background] Ananda P, Semedi BP, Waloejo CS, Utariani A. Opioid-Sparring and Multimodal Analgesia as Parts of Enhanced Recovery After Surgery (ERAS) Applied In The Ksatria Airlangga Floating Hospital. Indones J Anesthesiol Reanim 2021;3:17. https://doi.org/10.20473/ijar.v3i12021.17-21.
- [Background] Gramlich LM, Sheppard CE, Wasylak T, Gilmour LE, Ljungqvist O, Basualdo-Hammond C, Nelson G. Implementation of Enhanced Recovery After Surgery: a strategy to transform surgical care across a health system. Implement Sci. 2017 May 19;12(1):67. doi: 10.1186/s13012-017-0597-5. PMID 28526041
- [Background] Zychowicz A, Pisarska M, Laskawska A, Czyz M, Witowski J, Kisielewski M, Kulawik J, Budzynski A, Pedziwiatr M. Patients' opinions on enhanced recovery after surgery perioperative care principles: a questionnaire study. Wideochir Inne Tech Maloinwazyjne. 2019 Jan;14(1):27-37. doi: 10.5114/wiitm.2018.77261. Epub 2018 Jul 24. PMID 30766626
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Feng J, Li K, Xu R, Feng H, Han Q, Ye H, Li F. Association between compliance with enhanced recovery after surgery (ERAS) protocols and postoperative outcome in patients with primary liver cancer undergoing hepatic resection. J Cancer Res Clin Oncol. 2022 Nov;148(11):3047-3059. doi: 10.1007/s00432-021-03891-1. Epub 2022 Jan 25. PMID 35075571
- [Background] Rodriguez-Laiz GP, Melgar-Requena P, Alcazar-Lopez CF, Franco-Campello M, Villodre-Tudela C, Pascual-Bartolome S, Bellot-Garcia P, Rodriguez-Soler M, Miralles-Macia CF, Mas-Serrano P, Navarro-Martinez JA, Martinez-Adsuar FJ, Gomez-Salinas L, Jaime-Sanchez FA, Perdiguero-Gil M, Diaz-Cuevas M, Palazon-Azorin JM, Such-Ronda J, Lluis-Casajuana F, Ramia-Angel JM. Fast-Track Liver Transplantation: Six-year Prospective Cohort Study with an Enhanced Recovery After Surgery (ERAS) Protocol. World J Surg. 2021 May;45(5):1262-1271. doi: 10.1007/s00268-021-05963-2. Epub 2021 Feb 23. PMID 33620540
- [Background] Gillis C, Gill M, Marlett N, MacKean G, GermAnn K, Gilmour L, Nelson G, Wasylak T, Nguyen S, Araujo E, Zelinsky S, Gramlich L. Patients as partners in Enhanced Recovery After Surgery: A qualitative patient-led study. BMJ Open. 2017 Jun 24;7(6):e017002. doi: 10.1136/bmjopen-2017-017002. PMID 28647727